CLINICAL TRIAL: NCT05762913
Title: Effect of the Diaphragm Release Technique on Sleep Duration and Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Erkan Erol, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaU_Erol_07
Record Dates: First submitted 2023-02-19; First posted 2023-03-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Diaphragm; Relaxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diaphragm release (Experimental): The therapist passes his fingers under the costal arch, during inspiration the therapist accompanies the movement of the ribs, while during expiration he takes his fingers deeper, increasing his pressure. The therapist progresses progressively deeper into the costal arch with each breath. The maneuver will be performed in two sets of 10 deep breaths. The diaphragm release technique will be applied in 3 sessions, with 2 days of rest in between.
  Interventions: Other: Manual Diaphragm Release Technique

INTERVENTIONS:
Other: Manual Diaphragm Release Technique — The therapist passes his fingers under the costal arch, during inspiration the therapist accompanies the movement of the ribs, while during expiration he takes his fingers deeper, increasing his pressure. The therapist progresses progressively deeper into the costal arch with each breath. The maneuver will be performed in two sets of 10 deep breaths. The diaphragm release technique will be applied in 3 sessions, with 2 days of rest in between.

SUMMARY:
Even in healthy individuals, there may be tensions in the diaphragm muscle due to factors such as wrong posture, wrong breathing pattern, sedentary lifestyle, and it cannot fully fulfill its function. As a result of this tension in the diaphragm muscle, the breathing pattern deteriorates and sleep quality decreases. The aim of this study is to examine the effect of diaphragm release technique on sleep duration and sleep quality in healthy individuals. In this study, sleep quality of individuals will be evaluated with Pittsburgh Sleep Quality Index (PUKI), sleep duration, heart rate and step count with Fitbit® Inspire 2. 32 individuals living in Tokat will be included in the study. After obtaining the sociodemographic information of the individuals, the average of sleep duration, heart rate and step counts will be recorded for 3 days with the Fitbit® Inspire 2 wearable technology to be provided within the scope of the project. Sleep quality will be recorded with PUKI. The diaphragm release technique will be applied in 3 sessions, with 2 days of rest in between. After the applications are finished, sleep time, heart rate and step counts will be recorded for 3 days with Fitbit® Inspire 2 wearable technology.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65 who do not have any chronic disease or any past or present psychological disorder will be included.

Exclusion Criteria:

* Individuals with any neurological, psychiatric or cognitive impairment will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline
  In the scale consisting of 24 questions in total, 19 questions are answered by the person, while the other 5 questions are filled by the person's bedmate. 7 sub-dimensions (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are evaluated with 19 questions answered by the individual. Each item in the scale scores between 0 (no distress)-3 (severe distress). The sum of the scores of the seven sub-dimensions gives the total PSQI score (between 0-21). Those with a total score of 5≥ "good sleep", and those with a score of <5 are considered "poor sleep quality"
Pittsburgh Sleep Quality Index | 3rd day
  In the scale consisting of 24 questions in total, 19 questions are answered by the person, while the other 5 questions are filled by the person's bedmate. 7 sub-dimensions (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are evaluated with 19 questions answered by the individual. Each item in the scale scores between 0 (no distress)-3 (severe distress). The sum of the scores of the seven sub-dimensions gives the total PSQI score (between 0-21). Those with a total score of 5≥ "good sleep", and those with a score of <5 are considered "poor sleep quality"
Sleep Time | 3rd day
  Measurements will be made with the Fitbit® Inspire 2 device
Heart Rate | 3rd day
  Measurements will be made with the Fitbit® Inspire 2 device
Step Count | 3rd day
  Measurements will be made with the Fitbit® Inspire 2 device

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

REFERENCES:
- [Derived] Erol E, Kurtbogan M. The effects of diaphragm release on sleep quality: a pilot feasibility study. BMC Pulm Med. 2025 Oct 15;25(1):471. doi: 10.1186/s12890-025-03968-4. PMID 41094450